CLINICAL TRIAL: NCT05896618
Title: Evaluation of The Dental and Skeletal Effect of Transpalatal Arch and Nance Holding Arch as a Space Maintainers in Children: A Prospective Clinical Trial
Brief Title: Evaluation of Dental and Skeletal Effect of TPA and Nance as a Space Maintainers in Children: A Prospective Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Abd Elmajeed Omar Hussien, dentist, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TPA and Nance space maintainer
Record Dates: First submitted 2023-05-19; First posted 2023-06-09 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Dental Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): TPA group
  Interventions: Device: TPA
- Group II (Experimental): Nance group
  Interventions: Device: Nance appliance

INTERVENTIONS:
Device: TPA — 1. Group I (TPA group).In which patients will receive Transpalatal arch appliance as a space maintainer. Before treatment, dental cast will be made.Lateral cephalometric radiograph and extra-oral and intra-oral photographs will be taken for each patient. After 6 month follow up period, new cast will be made. New lateral cephalometric radiographs and new extra-oral and intra-oral photographs will be taken for each patient.
  Arms: Group I
Device: Nance appliance — 2. Group II (Nance group).In which patients will receive Nance holding arch appliance as a space maintainer. Before treatment, dental cast will be made.Lateral cephalometric radiograph and extra-oral and intra-oral photographs will be taken for each patient. After 6 month follow up period, new cast will be made. New lateral cephalometric radiographs and new extra-oral and intra-oral photographs will be taken for each patient.
  Arms: Group II

SUMMARY:
This study will aim to evaluate the dental and skeletal effect of the Transpalatal arch and Nance holding arch as a space maintainers in children.

DETAILED DESCRIPTION:
Primary teeth play a critical role in the growth and development of a child. In addition to their role in esthetics, eating, speech, and to encourage normal function and resultant expected growth, the other main function of a primary tooth is to hold space for the permanent successor until it is ready to erupt. The loss of multiple primary molars in the primary or mixed dentition can lead to many disturbances of the developing dentition and occlusion unless an appliance is constructed to maintain the relationship of the remaining teeth and to guide the eruption of the developing teeth. Space management is an important issue in pediatric dentistry, and many studies have been published about space maintainers related to the early extraction of primary teeth.

Several techniques have been used to protect the mesiodistal relationship of the teeth on the central arch. One of the best therapies is space maintainer therapy, because it could maintain those primary molars to be exfoliated naturally. The goals of the space maintainer treatment are to prevent teeth from drifting and reducing the space available for the permanent teeth, or to maintain some spaces within the arch so that alignment becomes possible. With the premature loss of a second primary molar, Nance holding arch or Transpalatal (TPA) appliance can be used on the maxillary arch and the lower lingual holding arch (LLHA) for the mandibular arch. The TPA is constructed from 0.9 or 1.25 mm stainless steel wire and crosses the palate to connect one molar or premolar to a contralateral tooth. This connection can be fixed by welding/soldering or be removable by insertion into a lingual sheath on the molar bands. These molar band sheaths are known as Wilson tubes or Mershon attachments. A modification of the attachment involves bonding the palatal wire directly to the lingual surface of the molars.

A modified maxillary lingual arch was described by Nance in 1947 and has since been commonly known as the Nance holding arch. The Nance appliance or Nance palatal arch (NPA) was one of the earliest modifications of the TPA. The palatal wire is welded/soldered to the molar bands and is connected anteriorly by an acrylic button positioned in the highest part of the palatal vault resting on non-compressible mucosa. The button is made of heat-cured, cold-cured or lightcured acrylic. Light-cured composite has also been used. Although the acrylic button can be very effective at resisting mesial drift, it does make it difficult for patients to maintain good oral hygiene due to the accumulation of food particles and plaque under the appliance. There is also the potential for tissue irritation and overgrowth of the tissues around the button.The dimensional changes are an important issue when we are interested in evaluation of Transpalatal arch and Nance holding arch. Dimensional changes include protrusion or intrusion of jaw as skeletal changes and proclination and retroclination of incisors as dental changes and also changes in arch length, arch width, intercanine distance and intermolar changes can be detected. Because of this, many studies have investigated arch dimensional changes in various stages of growth and development, such as arch width and arch dimensions. From the previous information that confirm that many problems may occur due to premature loss of maxillary primary molar without space maintainer appliance. Several studies investigate Transpalatal arch and Nance holding arch appliance, but no study interest to evaluate the dental and skeletal effect of both appliances. In this sense, this study will aim to assess the dental and skeletal effectiveness of Transpalatal arch and Nance holding arch appliance.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 9 years old.
* Skeletal class I or II
* Mixed dentition.
* The permanent incisors and primary canines were present in the maxillary arch.

Exclusion Criteria:

* Craniofacial anomalies.
* Skeletal posterior crossbite.
* Congenital missing teeth.
* Use of any space maintainer other than Transpalatal arch or Nance holding arch.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-03-05 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-06-08 (Estimated)

PRIMARY OUTCOMES:
Study cast and cephalometric measurements | 6 months
  - Lateral cephalograms measurements: At T1 (before treatment) and at T2 (after 6 month). Lateral cephalograms were traced digitally to measure the angles in degrees
  - Dental cast measurements: At T1 and T2. Study casts were made using alginate impressions to evaluate:
  1. Arch length in mm.
  2. Arch depth in mm
  3. Intermolar width in mm
  4. Intercanine width in mm

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Eldin Ismail, Study Chair — professor; Ahmed El awady, Study Director — lecturer; Hamdy Badreldin, Study Director — lecturer
Locations (2):
- Egypt (2):
  - Egypt, Cairo
  - Mahmoud Ahmed Abd Elmajeed Omar Hussien, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simon T, Nwabueze I, Oueis H, Stenger J. Space maintenance in the primary and mixed dentitions. J Mich Dent Assoc. 2012 Jan;94(1):38-40. PMID 22439522
- [Background] Raucci G, Pacheco-Pereira C, Grassia V, d'Apuzzo F, Flores-Mir C, Perillo L. Maxillary arch changes with transpalatal arch treatment followed by full fixed appliances. Angle Orthod. 2015 Jul;85(4):683-9. doi: 10.2319/070114-466.1. Epub 2014 Oct 6. PMID 25286341